CLINICAL TRIAL: NCT01071486
Title: Busulfan Pharmacokinetic Analysis and Glutathione S-transferase (GST)Genetic Polymorphism (A1,T1,M1,P1)in Adults Undergoing Hematological Bone Marrow Transplantation (HSCT).
Brief Title: Busulfan Pharmacokinetic Analysis and GST Polymorphism in Adults Undergoing Hematological Stem Cell Transplantation
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of participants
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Israel Cancer Association (Other)
Responsible Party: Principal Investigator, N_Krivoy, Clinical Pharmacology Unit, Rambam Health Care Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BU-AdultPK/PGx1
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Busulfan Pharmacokinetic Analysis; GST Genetic Polymorphism
Keywords: Busulfan; Glutathione S-transferase; Genetic polymorphism; HVOD; GVHD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Hematological Stem Cell Transplantation — Oral or Intravenous Busulfan as part of the preparative protocol for transplantation

SUMMARY:
Between 100 up to 200 adults undergoing HSCT for their primary disease will be included in this pharmacokinetic/pharmacogenetic study. In the preparative protocol Busulfan (BU)will be included as indicated in a known protocol. The GST polymorphism (A1,M1,T1 and P1) will be investigated using real time PCR. A correlation between pharmacokinetic parameters and patients polymorphism will be performed using known statistical technics for comparison. The aims of this study are, to correlate the demographic data, clinical presentation, clinical outcomes of the included individuals, the BU kinetics and the GST polymorphism and to establish an outcome "map" for those who receive HSCT for their primary disease.

ELIGIBILITY:
Inclusion Criteria:

* Malignant or Benign Diseases who need hematological stem cell transplantation as part of their treatment
* Busulfan should be part of the preparative protocol

Exclusion Criteria:

* Known sensitivity or allergy to Busulfan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Hepatic Veno-Occlusive Disease, Graft versus host disease | every week after HSCT up to 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel